CLINICAL TRIAL: NCT06903793
Title: Effects of Cervical Manipulation on Cervical Rotation Range of Motion and Shoulder Rotational Range of Motion and Strength in Overhead Athletes
Brief Title: Effects of Cervical Manipulation on Cervical Rotation Motion and Shoulder Rotational Motion and Strength in Overhead Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sacred Heart University (Other)
Responsible Party: Principal Investigator, Jason Grimes, PT, PhD, OCS, ATC, Associate Professor, Sacred Heart University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2025-216
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cervical Spine; Manipulation, Spinal; Shoulder; Overhead Athlete
Keywords: cervical manipulation; shoulder motion; shoulder strength; overhead athlete
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Masking Description: the researchers performing the pre- and post-intervention measures will be blinded to the results of those measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical manipulation (Experimental): All participants will be enrolled in the experimental group
  Interventions: Other: cervical manipulation

INTERVENTIONS:
Other: cervical manipulation — Cervical upglide/rotation manipulation targeted to C5/C6 on the dominant shoulder side

SUMMARY:
This study will examine the effects of a single session of a quick stretch technique delivered to the neck on neck and shoulder motion as well as shoulder strength in collegiate overhead athletes.

DETAILED DESCRIPTION:
Athletes participating in sports such as baseball, softball, tennis, swimming, and volleyball, are uniquely predisposed to cervical and shoulder dysfunction due to repetitive, high-intensity movements that require coordination between the cervical spine, shoulder, and upper extremities. These repetitive motions involve extreme glenohumeral (GH) range of motion (ROM) as well as high angular velocities, often leading to adaptations such as Glenohumeral Internal Rotation Deficit (GIRD). Overhead athletes with GIRD are at a higher risk of developing shoulder injuries.

This study aims to assess the effects of cervical spinal manipulation on cervical rotation ROM, GH rotational ROM and strength in overhead athletes. The current body of literature suggests an association between cervical rotation ROM deficits and arm injury risk in professional and collegiate-level baseball players. Restrictions in the cervical spine may alter neural and muscular pathways, potentially contributing to decreased shoulder ROM, compromised strength, and impaired performance. Given the complex interplay of cervical spine and shoulder function, understanding how cervical manipulation impacts the kinetic chain can play a vital role in developing shoulder rehabilitation and preventative programs for overhead athletes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* Current overhead college athlete
* No mental health considerations such as generalized anxiety disorder, PTSD, and schizophrenia

Exclusion Criteria:

* Upper extremity surgery in the last year
* Current shoulder pain
* Current neck pain
* Recent episodes of vertigo, dizziness, and migraines
* Recent motor vehicle accident
* History of cardiovascular disease such as hypertension, heart attack, stroke, coronary artery disease, peripheral artery disease, arrhythmias, heart valve disease, congenital heart defects, and aortic aneurysm
* Fear or unwillingness to undergo cervical manipulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Cervical rotation active range of motion | from baseline to immediately post-intervention
  Cervical rotation active ROM will be measured using the Cervical Range of Motion (CROM) device
Shoulder Rotational range of motion | from baseline to immediately post-intervention
  Dominant shoulder external rotation and internal rotation passive ROM at 90° of shoulder abduction will be measured using a digital inclinometer
Shoulder Rotational strength | from baseline to immediately post-intervention
  Dominant shoulder external rotation and internal rotation strength will be measured using the Hoggan MicroFET2 handheld dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Sacred Heart University, Fairfield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laudner KG, Stanek JM, Meister K. Assessing posterior shoulder contracture: the reliability and validity of measuring glenohumeral joint horizontal adduction. J Athl Train. 2006 Oct-Dec;41(4):375-80. PMID 17273461
- [Background] Keller RA, De Giacomo AF, Neumann JA, Limpisvasti O, Tibone JE. Glenohumeral Internal Rotation Deficit and Risk of Upper Extremity Injury in Overhead Athletes: A Meta-Analysis and Systematic Review. Sports Health. 2018 Mar/Apr;10(2):125-132. doi: 10.1177/1941738118756577. Epub 2018 Jan 30. PMID 29381423
- [Background] Bullock GS, Thigpen CA, Zhao H, Devaney L, Kline D, Noonan TJ, Kissenberth MJ, Shanley E. Neck range of motion prognostic factors in association with shoulder and elbow injuries in professional baseball pitchers. J Shoulder Elbow Surg. 2025 Feb;34(2):421-429. doi: 10.1016/j.jse.2024.08.026. Epub 2024 Oct 11. PMID 39396612
- [Background] Devaney LL, Denegar CR, Thigpen CA, Lepley AS, Edgar C, DiStefano LJ. Preseason Neck Mobility Is Associated With Throwing-Related Shoulder and Elbow Injuries, Pain, and Disability in College Baseball Pitchers. Orthop J Sports Med. 2020 May 18;8(5):2325967120920556. doi: 10.1177/2325967120920556. eCollection 2020 May. PMID 32523967
- [Background] Cools AM, De Wilde L, Van Tongel A, Ceyssens C, Ryckewaert R, Cambier DC. Measuring shoulder external and internal rotation strength and range of motion: comprehensive intra-rater and inter-rater reliability study of several testing protocols. J Shoulder Elbow Surg. 2014 Oct;23(10):1454-61. doi: 10.1016/j.jse.2014.01.006. Epub 2014 Apr 13. PMID 24726484